CLINICAL TRIAL: NCT06490393
Title: The Impact of Supervision by a Health Care Professional on Quality of Life (QoL) Questionnaire Scoring and Completion:, Randomized, Cross-over Study in Cancer Patients Receiving Systemic Antineoplastic Therapy
Brief Title: The Impact of Supervision by a Health Care Professional on Quality of Life Questionnaire
Acronym: IMSUP
Status: Recruiting | Type: Observational
Sponsor: St. Claraspital AG (Other)
Responsible Party: Principal Investigator, Diana de Jong, Principal Investigator, St. Claraspital AG
Other Study IDs: IMSUP
Record Dates: First submitted 2024-06-04; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Health-related Quality of Life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A:paper vs digitally: Arm A: patients in Arm A will receive first an invitation to complete the QoL questionnaires on paper under supervision of an HCP in the hospital before their cycle of systemic antineoplastic therapy starts. Prior to their subsequent cycle of systemic antineoplastic therapy (regardless of duration of cycle), patients in Arm A will be asked to complete the same QoL questionnaires digitally at home.
  Interventions: Other: Questionnaires
- B: digitally vs paper: Arm B: patients in Arm B will receive first an invitation to complete the QoL questionnaires digitally at home before their cycle of systemic antineoplastic therapy starts. Prior to their subsequent cycle of systemic antineoplastic therapy (regardless of duration of cycle), patients in Arm B will be asked to complete the same QoL questionnaires on paper under supervision in the hospital.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — EORTC QLQ-C30 (General Health), EORTC QLQ-SH22(sexual Health), Financial questionnaire as routinely used by the Social Department

SUMMARY:
Effect of supervision on scoring and completion on Quality of Life Questionnaire

DETAILED DESCRIPTION:
This protocol will study the impact of supervision on completion and scoring of sensitives domains of QoL Questionnaires and QoL Questionnaires in general in a multi-center, randomized, cross-over design in cancer patients receiving systemic antineoplastic therapy

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age and legally competent
* Signed informed consent available
* Systemic oncologic treatment (e.g. chemotherapy, immunotherapy, endocrine therapy)
* Current systemic therapy started at least 4 weeks before randomization and is scheduled to continue for at least another 4 weeks after randomization in the same dose and interval
* Patient is ready and able to complete quality of life questionnaires in German (on paper

Exclusion Criteria:

* One or more of the inclusion criteria not met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to enroll at least 200 patients into this study. Patient recruitment will be conducted during 2 years (2024-2026)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | 2024-2026
  To study the impact of Health Care Professional supervision on scoring patterns on financially- and sexuality related questions by cancer patients receiving systemic antineoplastic therapy, compared to self-administered electronic completion at home. The null-hypothesis is tested that the method of administration does not influence patients' answers.
EORTC QLQ-SH22 | 2024-2026
  To study the impact of Health Care Professional supervision on scoring patterns on financially- and sexuality related questions by cancer patients receiving systemic antineoplastic therapy, compared to self-administered electronic completion at home. The null-hypothesis is tested that the method of administration does not influence patients' answers.
Questionnaire called "Financial consequences" routinely used by the Social department of St. ClaraSpital | 2024-2026
  To study the impact of Health Care Professional supervision on scoring patterns on financially- and sexuality related questions by cancer patients receiving systemic antineoplastic therapy, compared to self-administered electronic completion at home. The null-hypothesis is tested that the method of administration does not influence patients' answers.

SECONDARY OUTCOMES:
Incidence of reported sexual problems | 2024-2026
Patient preference | 2024-2026
  Reported patient preference of mode of reporting (electronically vs supervised)
Time | 2024-2026
  Time used by the Health care professional per completion mode

CONTACTS AND LOCATIONS:
Overall Officials: Diana de Jong-Bakker, Principal Investigator — St. Claraspital Klinische Forschung
Locations (1):
- St Clara Research Ltd, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No